CLINICAL TRIAL: NCT06150105
Title: Changes in the Hormonal and Inflammatory Profile of Young Sprint- and Endurance-trained Athletes Following a Sports Camp
Brief Title: Changes in the Hormonal and Inflammatory Profile of Young Sprint- and Endurance-trained Athletes.
Acronym: CHIPYA
Status: Completed | Type: Observational
Sponsor: Poznan University of Physical Education (Other)
Responsible Party: Sponsor
Other Study IDs: 530/18
Record Dates: First submitted 2023-11-13; First posted 2023-11-29 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-11

CONDITIONS: Overtraining Syndrome
Keywords: epinephrine, norepinephrine, cortisol, athletes, fatigue
MeSH Terms: conditions — Overtraining Syndrome; Fatigue | interventions — Exercise

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- sprint-trained: Sprint-trained athletes: 6 male and 6 female, aged average 15 y.,
  Interventions: Other: Exercise training
- endurance-trained: Endurance-trained athletes: 6 male and 6 female, aged average 15 y.,
  Interventions: Other: Exercise training

INTERVENTIONS:
Other: Exercise training — Intense endurance training

SUMMARY:
One essential element of athlete training is conditioning camps, where athletes undergo a rigorous and targeted training schedule to prepare for upcoming sporting events. During sports camps, due to the accumulation of a large number of training units, including high-intensity exercises, athletes react with post-exercise overload, acute fatigue, and overreaching which can become a chronic overtraining syndrome. Overtraining syndrome is a very specific and severe condition where overtraining without adequate rest and recovery leads to performance decrements lasting more than 2-3 months, coupled with a mood disturbance. The exact etiology and pathogenesis are unknown and actively being investigated.

During training camps the balance between training volumes and recovery is often a delicate one and, the accumulation of exercise-induced stress may exceed the capacity of both neuroendocrine and immune adaptation leading to an alteration of physiological functions, decreasing adaptation to performance, impairment of psychological processing, immunological dysfunction, and biochemical abnormalities. Moreover, there is currently a lack of biomarkers accessible to assist in diagnosing and, what's even more important - help to prevent the overtraining syndrome, except for the continued presence of unexplained underperformance despite athletes' adequate rest and recovery.

Thus, this study aims to explain how long and intensive training for endurance affects the hormonal and immune systems of young athletes.

The main questions it aims to answer are:

1. How does intense training influence hormonal and immune responses in young, trained athletes?
2. Does training specialization affect the hormonal and immune response to intense training?

DETAILED DESCRIPTION:
Twenty-four young male and female athletes, specializing in athletics disciplines such as sprint (hurdles, 100m, 110m), and endurance: race walk, 5000m, and 10000m, volunteered to take part in this study. Investigation was held during 9 days of the training camp (preparatory period, general preparation sub-period), which was aimed at increasing the endurance and flexibility of athletes. During the training camp, all subjects occupied the same accommodations and followed the same training plan and diet schedules. The camp regime included 2 training sessions per day, lasting 4 hours per day, and a total of 21 hours per 9 days. Blood samples were taken always in the same conditions, from the antecubital veins. Participants were seated in a recumbent position for a minimum of 10 minutes before blood draws to stabilize the hydrostatic condition. Before collection of the first sample (rested baseline), participants were asked to avoid any intense exercise at least 24 hours before sampling. Next samples were taken after 4 days and after another 5 days of training camp (in total after 9 days). The concentration of catecholamines: epinephrine and norepinephrine in serum was measured as well and the responsiveness of the adrenal medulla to the sympathetic nervous activity was estimated by the ratio E/NE calculated. Also, concentrations of cortisol, hs-CRP, and myoglobin were measured and changes in blood morphology were estimated.

ELIGIBILITY:
Inclusion Criteria:

* age 15-17 years,
* minimum of 3 years of training experience,
* specialization in anaerobic and aerobic disciplines.

Exclusion Criteria:

* presence of acute or chronic inflammation
* fever, infections, injuries
* se of any anti-inflammatory drugs.

Ages: 15 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Twenty-four young male and female athletes, students at Sports Championship School, future representatives of the Polish National Team, specializing in athletics disciplines such as sprint (hurdles, 100m, 110m), and endurance: race walk, 5000m, and 10000m, volunteered to take part in this study.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2018-02-16 (Actual); Primary Completion 2018-02-24 (Actual); Study Completion 2018-12-10 (Actual)

PRIMARY OUTCOMES:
Changes in epinephrine serum level. | at rest baseline (before training), after 4 - and after another 5 days of training.
  marker of HPA axis functioning, stress hormone.
Changes in norepinephrine serum level. | at rested baseline (before training), after 4 - and after another 5 days of training.
  marker of HPA axis functioning, stress hormone.
Changes in cortisol serum level. | at rested baseline (before training), after 4 - and after another 5 days of training.
  marker of HPA axis functioning, stress hormone
Changes in hs-CRP serum level. | at rested baseline (before training), after 4 - and after another 5 days of training.
  marker of inflammatory response.
Changes in Myoglobin serum level. | at rested baseline (before training), after 4 - and after another 5 days of training.
  marker of muscle damage

SECONDARY OUTCOMES:
Changes in blood morphology. | sat rested baseline (before training), after 4 - and after another 5 days of training.
  Morphometric measurements of blood cell.
Changes in epinephrine/norepinephrine ratio. | at rested baseline (before training), after 4 - and after another 5 days of training.
  marker of responsiveness of the adrenal medulla to sympathetic nervous activity.

CONTACTS AND LOCATIONS:
Overall Officials: Joanna Ostapiuk-Karolczuk, Ph.D., Principal Investigator — Poznan University of Physical Education
Locations (1):
- Poznań University of Physical Education, Poznan, Poland

REFERENCES:
- [Derived] Ostapiuk-Karolczuk J, Kasperska A, Dziewiecka H, Cieslicka M, Zawadka-Kunikowska M, Zaleska-Posmyk I. Changes in the hormonal and inflammatory profile of young sprint- and endurance-trained athletes following a sports camp: a nonrandomized pretest-posttest study. BMC Sports Sci Med Rehabil. 2024 Jun 20;16(1):136. doi: 10.1186/s13102-024-00924-3. PMID 38898468